CLINICAL TRIAL: NCT05251168
Title: Role of FDG PET/CT Guided Bone Marrow Biopsy vs. Conventional Bone Marrow Trephine Biopsy for Assessing the Bone Marrow Infiltration in Newly Diagnosed Lymphoma
Brief Title: PET Guided Bone Marrow Biopsy vs Trephine Bone Marrow Biopsy
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajender Kumar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: INT/IEC/2017/1416
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Lymphoma; Bone Marrow Neoplasm
MeSH Terms: conditions — Lymphoma; Bone Marrow Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PET Guided Bone Marrow Biopsy — The results of PET/CT images were discussed with the referring physician. PET/CT targeted metabolic marrow biopsy was planned two hours after the whole body diagnostic imaging or on a subsequent day one hour after injecting 2-3 mCi of FDG to minimize the radiation exposure burden to the interventionist.
  Society of Interventional Consensus guidelines was followed for image-guided biopsy.
  The bone marrow biopsy was done under the PET/CT guidance using the same PET/CT scanner with the help of an automated robotic arm (ARA) workstation
Procedure: Trephine Bone Marrow Biopsy — All the participants underwent trephine bone marrow biopsies from the bilateral posterior superior iliac spine before treatment planning.

SUMMARY:
Newly diagnosed lymphoma patients were recruited for FDG PET/CT and PET/CT guided bone marrow biopsy. All the patients also underwent routine bone marrow sampling from the posterior superior iliac spine.

DETAILED DESCRIPTION:
Newly diagnosed patients underwent FDG PET/CT for whole-body staging. All the PET/CT images were analyzed by a qualified nuclear medicine physician. The bone marrow FDG uptake was classified as negative, focal, multifocal and diffuse marrow uptake. A PET/CT guided metabolic bone marrow sampling from the FDG avid marrow-based lesion was done. However, patients with diffuse FDG avidity or no uptake in the marrow differed for PET-guided biopsy. All the patients underwent routine trephine bone marrow sampling. Bone marrow infiltration (final diagnosis) was established based on trephine bone marrow sampling and FDG PET/CT targeted bone marrow biopsy results in the present study. The results of both the biopsies were correlated with the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed cases of lymphoma (both HL and NHL).
2. Hypermetabolic bone marrow lesions on staging 18F-FDG PET/CT, which are accessible for biopsy.
3. Aged between 18 -80 years.
4. Informed consent prior to the procedure.

Exclusion Criteria:

1. Previously treated/relapsed lymphoma.
2. Initiation of therapy (chemotherapy, radiation therapy) and/or hematopoietic growth factor injections before 18F-FDG PET/CT or BMTB.
3. Patients who underwent a prior BMTB to evaluate the role of BMI.
4. Patients with pre-existing bleeding diatheses like hemophilia, coagulopathy, INR > 1.2 and platelet counts < 50,000/mm3,
5. Patients who refuse to provide informed consent.
6. No 18F FDG avid skeletal lesions.
7. Pregnant/Lactating female patients.
8. Non-cooperative patients.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Treatment naïve patients of lymphoma who underwent FDG PET/CT for initial staging were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison results of PET guided bone marrow biopsy with trephine bone marrow biopsy | three months
  The final diagnosis of bone marrow infiltration was based on the pathology findings of trephine bone marrow biopsy and FDG PET/CT targeted bone marrow biopsy.
  The diagnostic accuracy (in percentage) of FDG PET/CT guided metabolic bone marrow biopsy was compared with the accuracy (in percentage) of trephine bone marrow biopsy with respect to final diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
Study protocol can be shared only on reasonable requests.